CLINICAL TRIAL: NCT04512417
Title: A Multi-Center, Randomized Controlled, Phase II Clinical Study Of Camrelizumab With Or Without Radiotherapy For The Treatment Of Recurrent Or Metastatic Esophageal Cancer That Has Progressed After Chemotherapy
Brief Title: A Clinical Study Of Camrelizumab With Or Without Radiotherapy In The Treatment Of Esophageal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB-2020-176
Record Dates: First submitted 2020-08-11; First posted 2020-08-13 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Esophageal Cancer
Keywords: Esophageal Cancer; Camrelizumab; IO、Radiotherapy
MeSH Terms: conditions — Esophageal Neoplasms | interventions — camrelizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined radiotherapy group (Experimental)
  Interventions: Drug: Camrelizumab+Radiotherapy
- Immunotherapy alone group (Experimental)
  Interventions: Drug: Camrelizumab

INTERVENTIONS:
Drug: Camrelizumab+Radiotherapy — The combined treatment group received radiotherapy for recurring or metastatic lesions: at least one or more lesions were irradiated, stereotactic body radiotherapy (SBRT, 8Gy/time, 3-5 times) or conventional radiotherapy (parts not suitable for SBRT, total Dose 30Gy or more); start immunotherapy within 8 weeks after radiotherapy.Until PD or toxicity is intolerable or up to 24 months.
  Other Names: SBRT
  Arms: Combined radiotherapy group
Drug: Camrelizumab — Camrelizumab,200mg,Q3W,Until PD or toxicity is intolerable or up to 24 months.
  Arms: Immunotherapy alone group

SUMMARY:
The purpose of this study is to observe and evaluate the efficacy and safety of Camrelizumab combined with or without radiotherapy for the treatment of recurrent or metastatic esophageal cancer that has progressed after chemotherapy

DETAILED DESCRIPTION:
In China, the incidence of esophageal cancer has declined in recent years, but the mortality rate has been ranked fourth. Morbidity and mortality were ranked sixth and fourth in all malignancies, respectively. Therefore, esophageal cancer has always been a major malignant tumor that threatens the health of our residents. We designed a multi-center, randomized controlled, phase II clinical study of camrelizumab with or without radiotherapy for the treatment of recurrent or metastatic esophageal cancer that has progressed after chemotherapy. The purpose of this study is to observe and evaluate the efficacy and safety of camrelizumab with or without radiotherapy for advanced esophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

* 1. Volunteer to participate in clinical research: fully understand and know the research and sign the Informed Consent Form (ICF); willing to follow and have the ability to complete all trial procedures;
* 2. Recurrent or metastatic esophageal cancer confirmed by histology or cytology, patients with ≤4 metastatic lesions;
* 3. Progress after first-line chemotherapy;
* 4. There are lesions measurable according to RECIST standards
* 5. Age ≥18 years old and ≤75 years old, regardless of gender
* 6. ECOG physical strength status score is 0～2;
* 7. Have not received immunotherapy or biological therapy before;
* 8. Hemoglobin ≥90g/L, platelets ≥10×109/L, absolute neutrophil count ≥1.5×109/L;
* 9. Serum creatinine ≤1.25 times UNL or creatinine clearance ≥60 mL/min;
* 10. Serum bilirubin≤1.5×UNL, AST (SGOT) and ALT (SGPT)≤2.5×UNL, alkaline phosphatase≤5×UNL;
* 11. No history of interstitial pneumonia or previous interstitial pneumonia;

Exclusion Criteria:

* 1. Previously received anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137 or anti-CTLA-4 antibody treatment, or any other antibodies targeting T cell costimulation or checkpoint pathways as specific targets or drug;
* 2. Have received radiotherapy in the past, and the tumor in the irradiation field has progressed;
* 3. Metastasis of meninges, pleura or pericardium;
* 4. Esophageal perforation and active esophageal bleeding, with invasion of trachea and large blood vessels in the thoracic cavity;
* 5. Patients with severe cardiovascular or pulmonary diseases, interstitial pneumonia or previous history of interstitial pneumonia:
* 6. Patients who cannot understand the test requirements or may not comply with the test requirements;
* 7. Autoimmune diseases (such as: systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, autoimmune thyroid disease), but allow the following diseases to enter the next step of screening: type I diabetes, skin that does not require systemic treatment Diseases (such as vitiligo, psoriasis);
* 8. Active hepatitis B or C that requires treatment;
* 9. Suffered from an active infection requiring systemic treatment 14 days before the first administration;
* 10. Patients with other malignant lesions, except for curable skin cancer (non-melanoma), cervical carcinoma in situ or malignant disease cured ≥5 years;
* 11. The researcher believes that some obvious diseases should be excluded from this research;
* 12. The dose limit of radiotherapy cannot meet the limit requirement set by this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2020-08-31 (Estimated); Primary Completion 2021-08-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) per RECIST 1.1 | Up to 24 months
  PFS is defined as the time from randomization to the first documented disease progression per RECIST 1.1 based on blinded independent central review or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 | Up to approximately 6 months.
  ORR is defined as the percentage of participants in the analysis population who have a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: ≥30% decrease in the sum of diameters of target lesions) per RECIST 1.1.
Overall Survival (OS) | Up to 24 months
  defined as the time from randomization to death from any cause during the course of the study.
Number of Subjects with treatment-related adverse events (AEs) | Up to 24 months
  Incidence, nature, and severity of adverse events graded according to the NCI CTCAE v5.0.
Failure mode | Up to 24 months
  Observe and collect the reasons for the treatment failure of the subjects during the study

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Province Cancer Hospital, Hanzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided